CLINICAL TRIAL: NCT00336752
Title: A Prospective Randomized Multi-Centre Study to Compare Operative Versus Non Operative Functional Treatment in Patients With Unstable Isolated Fibula Fractures
Brief Title: Operative Versus Non Operative Treatment for Unstable Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Sanders, Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-03-113; HSREB09641 (Other: Western University Research Ethics)
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Ankle Injuries
Keywords: undisplaced ,unstable wEBER B ankle fractures; operative intervention; non operative intervention
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Non operative treatment of Weber B ankle fracture. Use of cast, with no surgical intervention
  Interventions: Procedure: non operative treatment
- 2 (Active Comparator): Operative treatment of Weber B ankle fracture. Open reduction and internal fixation to repair a broken bones.
  Interventions: Procedure: operative treatment of ankle fractures

INTERVENTIONS:
Procedure: non operative treatment — non operative treatment -casting for 6 weeks
  Arms: 1
Procedure: operative treatment of ankle fractures — operative treatment of ankle fractures
  Arms: 2

SUMMARY:
The purpose of the study is to compare functional outcomes and recovery following surgical and non surgical treatment of potentially unstable , isolated fibula fractures. Secondary objectives are to compare the re-operation rate, time to union and complications between the two treatment groups.

The primary research questions:

1. Does surgery provide a better functional outcome compared to non operative treatment of undisplaced, unstable fractures?
2. Do patients with these fractures return to activities faster after operative or non operative treatment?
3. Are complications more common with operative or non operative care?

DETAILED DESCRIPTION:
The most controversial ankle fracture is the Weber B fracture in which the fibular (or lateral malleolar) fracture begins at the level of the ankle mortise and extends proximal and lateral. This fracture can exist as isolated fractures of the lateral malleolus, or bimalleolar injuries in which both lateral and medial malleoli are fractured. When both malleoli are fractured, the ankle has lost all of its bony support and is unstable. In contrast, if only the lateral malleolus is injured, the Weber B injury may be either stable or unstable. When the ankle is subluxed or dislocated in these injuries, the ankle is clearly unstable. However, when the ankle is not initially subluxed, the assessment of stability is more difficult. Stability in isolated lateral malleolar fractures depends upon the status of the medial, or deltoid, ligaments. Further complicating matters, the deltoid ligament may be intact, partially torn, or completely torn such that there is a spectrum of stability for these injuries.Previous studies relied upon an assessment of tenderness over the ligament to determine instability, but this may not differentiate between partial and complete tears.

In North America, most surgeons would agree that markedly unstable definitely unstable ankle fractures are best treated surgically.Therefore, Weber B fractures which involve fractures of both the medial and lateral malleolus are best treated by surgical stabilization. Furthermore, Weber B fractures involving only the lateral malleolus, but which present with lateral subluxation of the talus, are definitely unstable and require fixation.

In contrast, controversy exists between surgeons regarding the optimal means of treating an undisplaced but potentially unstable fibula fracture. Many surgeons recommend routine operative fixation, while others recommend routine non-operative treatment.A clear rationale exists for both types of treatment.

The most important factor in treatment includes maintaining the reduction of the talus within the ankle mortise. Even 1 mm of displacement or lateral shift of the talus will affect ankle joint loading and lead to dysfunction and potentially arthritis. Other issues include the potential benefits of earlier mobilization and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature male or female < 65 years of age
2. Unstable ankle on stress exam: medial clear space ³ 5 mm: no Mortise shift on static radiographs
3. Unilateral Weber B fibular fractures
4. Closed fracture
5. Provision of informed consent -

Exclusion Criteria:

1. Fractures not amenable to surgical treatment
2. Pathologic fracture
3. Associated injuries to the foot, ankle, tibia, or knee
4. Associated medial malleolus fracture
5. Surgical delay of >2 weeks from time of injury
6. Previous fracture or retained hardware in the affected limb
7. Associated neurovascular injury or deficit in the affected limb
8. Systemic diseases including diabetes, multiple sclerosis, Parkinson's disease, and other disorders which might affect peripheral sensorimotor function -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome: comparison of physical functioning score on SF36 | enrolment, 6 weeks, 3,6 12 months

SECONDARY OUTCOMES:
Secondary objectives are to compare the re-operation rate between operative and non-operative treatment and to compare the time to union, rates of nonunion and complications such as infection between the two groups. | enrolment, 6 weeks, 3,6,12 months
  Number of participants with complications or adverse events that ae related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: DR. David Sanders, M.D., FRCSC, Principal Investigator — Western University, Canada
Locations (1):
- LOndon Health Sciences cEntre- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No